CLINICAL TRIAL: NCT05904639
Title: Multivariable Transcriptomic Analysis, Dietary Patterns and Cardiovascular Risk in African Americans
Brief Title: Decoding Your Diet (DYD)
Acronym: DYD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Morehouse School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1992237-3
Record Dates: First submitted 2023-05-08; First posted 2023-06-15 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Cardiovascular Disease
Keywords: diet; transcriptomics; gene expression; cardiovascular
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: In this study, we will implement a high quality AHA plant-based diet intervention on cardiac patients and study its effects on GE. We will use a GE-whole genome sequencing (WGS) cluster approach in which we will integrate genetic-biological technologies within pathways associated with CVD to create risk score clusters. We will develop risk scores and identify top (most significant by p value) genetic clusters in common functional pathways. We will further integrate genetic information with clinical factors and CVD risk factors and investigate association with AHA diet.
Who Masked: Participant
Masking Description: masking of participants to biostatistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pre-study (Experimental): Baseline or pre-study arm
  Interventions: Genetic: Decoding Your Diet
- Cross-over arm (Experimental): Intervention arm
  Interventions: Genetic: Decoding Your Diet

INTERVENTIONS:
Genetic: Decoding Your Diet — We will collect information from cardiac patients on their genes at baseline and then expose them to a diet intervention and collect genetic information after the intervention.

SUMMARY:
Our study will determine if a high quality AHA plant-based diet intervention can promote a genetic signature that is protective against CVD. Our development of GE mutational signatures in Blacks/African Americans with a high CVD burden can inform of changes patients can implement in their diet and lifestyle to decrease the CVD risk burden.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the US and worldwide, contributing to 1 in every 4 deaths. Compared to European Americans, African Americans have higher risks for cardiometabolic conditions. Our study aim is to determine if a high-quality American Heart Association (AHA) plant-based diet intervention can promote a genetic mutational signature that is protective against CVD. We will enroll 15 Black/African American cardiac patients from Grady Memorial Hospital, Atlanta, GA. We will investigate from baseline to 3 months how the AHA plant-based diet intervention affected the regulation of several genes that are differentially expressed (DEG) and cluster together within biological pathways. We will integrate this information with WGS data, clinical factors, and ASA24-hour recalls. We expect that the AHA plant-based diet will be protective against deleterious DEG patterns that promote development of CVD. Our DEG mutational signatures in Black/African Americans with a high CVD burden can inform of changes patients can implement in their diet to decrease CVD risk burden. Our study will also fill gaps in providing new information regarding novel genomic-biological signatures with diet predictors and risk factors of CVD that can be useful in designing prevention and treatment strategies in precision medical care.

ELIGIBILITY:
Inclusion Criteria

* Black or African American
* Age ≥ 40 years
* All sexes as determine by biology (sex chromosomes)
* ≥3 abnormal metabolic traits including diagnosed cardiometabolic diseases:
* At least Class I Obesity (BMI ≥ 30 kg/m2)
* High waist circumference: > 40 inches (102 cm) for men and > 35 inches (88 cm) for women
* Diagnosed cardiometabolic diseases or metabolic traits:
* diagnosed heart disease, stroke
* Peripheral vascular disease, carotid artery disease, type 2 diabetes without disability
* HbA1c > 6.4%, or fasting: >126 mg/dL or postprandial > 200 mg/dL or OGTT > 200 mg/dL
* ≥ grade 1 hypertension: SBP >140mmHg or dbp: > 90mmHg
* Triglycerides > 150mg/Dl
* Total cholesterol > 200 mg/dL
* HDL cholesterol <40 mg/dL for men or < 50 mg/dL for women
* LDL > 160 mg/dL; VLDL > 30 mg/dL

Exclusion Criteria:

* All other racial groups
* Age < 40 years
* Normal weight (BMI 18.5-24.9 kg/m2)
* Normal waist circumference < 40 inches (<102 cm) for men and < 35 inches (<88 cm) for women
* < 3 abnormal metabolic traits/ diagnosed cardiometabolic diseases
* Orthopedic conditions (i.e., recent hip or knee replacement)
* Paralysis
* Diagnosed severe dementia
* End-stage renal disease: chronic kidney disease: stage 3 or 4
* Congestive heart failure (advanced stage and not fluid-stable)
* Chronic fluid retention

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Differential changes in gene expression from baseline to end of study. | 3 months
  Differential changes in gene expression will be assessed by statistics. These changes will be assessed in response to changes in cardiovascular risk factors when the participants use an AHA plant-based diet.

CONTACTS AND LOCATIONS:
Locations (1):
- Morehouse School of Medicine, Atlanta, Georgia, United States